CLINICAL TRIAL: NCT03997864
Title: Administration of Prazosin to Prevent PTSD After Sexual Assault
Brief Title: Administration of Prazosin to Prevent PTSD in Adult Women After Sexual Assault
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID recruitment issues
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19-0733
Record Dates: First submitted 2019-06-20; First posted 2019-06-25 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Sexual Assault; Trauma; prevention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Prazosin

STUDY DESIGN:
Intervention Model Description: Participants in this study will include 40 adult females who complete consent (20 per arm), ages 18-50 years, who are evaluated and treated at the University of Colorado Hospital after an alleged sexual assault on their person. Randomization will be completed by the pharmacy and study condition (prazosin/treatment vs. placebo/control) masked throughout the data collection portion of the study. Participants will attend weekly visits during the 3-week medication trial and 2-3 week tapering off of medication, followed regular check-in phone calls with study staff between stopping the medication and the follow-up assessments at the final study visit (approx. 3 moths post study enrollment).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized double-blind placebo-controlled trial. All study team personnel (PI, RAs) and study participants will be blinded to intervention condition [prazosin (treatment) vs. placebo (control)] throughout active data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment - prazosin (Active Comparator): Participants randomized to this group will receive the medication prazosin.
  Interventions: Drug: Prazosin
- Control - placebo (Placebo Comparator): Participants randomized to this group will receive placebo .
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Prazosin — Starting dose: 2mg at HS. Maximum dose: 15 mg at HS. Dosage will be increased 1 mg every 3 days until sleep is improved, max dose is reached, or side effects are problematic.
  Tapering Decrease prazosin 1 mg every 3 days or 3 mgs per week until off completely. Tapering will take approximately 2-3 weeks.
  Other Names: Minipress
  Arms: Treatment - prazosin
Drug: Placebos — Starting dose: 2mg at HS. Maximum dose: 15 mg at HS. Dosage will be increased 1 mg every 3 days until sleep is improved max dose is reached, or side effects are problematic.
  Arms: Control - placebo

SUMMARY:
This study plans to learn more about whether taking the medication, Prazosin, immediately and during the weeks immediately following a traumatic event can help to reduce the risk of developing posttraumatic stress disorder (PTSD). Early post traumatic event sleep disturbance predicts the later development of PTSD. Prazosin has shown some effectiveness in reducing trauma related nightmares and sleep disturbance. We hypothesize that regulating sleep immediately after a sexual assault will reduce PTSD and diminish symptoms.

DETAILED DESCRIPTION:
This study plans to learn more about whether taking the medication, Prazosin, in the weeks immediately following a traumatic event can help to reduce the risk of developing posttraumatic stress disorder (PTSD).

Specific Aim 1: Test the efficacy of the drug prazosin in decreasing PTSD symptom severity as compared to placebo at 3 months post rape as measured by the Clinician-Administered PTSD Scale version 5 (CAPS-5, primary outcome) as well as associated secondary outcomes (PTSD diagnosis rate, sleep scores, and depression symptoms) at 3 months.

Hypotheses:

1a: Severity score on the CAPS-5 will be significantly lower in rape victims randomized to receive prazosin within 24 hours of at the University of Colorado Hospital (UCH) Emergency Department and continue on a titrated dose for one month compared to the control group at 3 months post rape. Secondarily, PTSD diagnosis rate will be lower in the prazosin group versus the control group at 3 months.

1b: Participants randomized to receive prazosin will have better sleep scores as measured by the Pittsburgh Sleep Quality Index (PSQI) and PSQI Trauma addendum at 3 months post rape as compared to the control group.

1c: Severity scores for major depressive symptoms as measured by the Patient Health Questionnaire (PHQ-9) will be significantly lower in rape victims randomized to receive prazosin as compared to the control group at 3 months post rape.

1d: Sleep scores as measured by the PSQI and PSQI Trauma addendum will be positively correlated with PTSD symptom severity as measured by the CAPS-5 such that higher (worse) sleep scores are associated with more PTSD symptoms.

Rationale: Many studies have shown that sleep disturbances and nightmares that occur directly after a traumatic event are a good predictor of the development of PTSD. Prazosin has been shown to improve PTSD-related sleep disturbance, including nightmares. If prazosin can effectively treat sleep disturbance in the weeks immediately following a traumatic experience and decrease the rate of PTSD and the severity of symptoms, then it could possibly become the standard of care for individuals exposed to a traumatizing event.

Brief overview of methods: Females between the ages of 18 and 50 years will be recruited directly from the ED at University of Colorado Hospital with the assistance of the Forensic Nurse Examiners. Those who elect to take part in this study and complete the informed consent process will be randomized to receive either prazosin or placebo. This is a double-blind study, so neither the participant nor the study doctor/team will know whether a participant is in the treatment (prazosin) or control (placebo) group. Participants will receive three 2mg tabs and three 1mg tbs for titration purposes (prazosin or placebo equivalent) before they leave the hospital, with instructions to take the first dose (2 mg) 1 hour before bed, the first night after being seen in the ED. Study staff will follow up the next day to inquire about the participant's general condition, possible side-effects, sleep, and to schedule the first study visit (at ~72 hours after treatment in ED). PTSD and posttraumatic stress symptoms, symptoms of depression, suicidality, medication compliance, side-effects and adverse events will be monitored and assessed by study personnel at weekly study visits for the duration of the med trial (~6 weeks; 3 weeks on medication and 2-3 weeks of tapering off of medication) and again at 3-months post. However, participants will be instructed to report any changes or concerns as needed. Each participant will also complete a daily sleep log for the duration of their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between the ages of 18 years and 50 years
* Victim of sexual assault/rape
* Able to understand consent procedure
* Discharged to home

Exclusion Criteria:

* Admitted to inpatient unit
* Previous diagnosis of PTSD
* Contra-indications to prazosin: orthostatic hypotension, right heart failure, use of anti-hypertensive medication, 5-phosphodiesterase inhibitors (sildenafil) or diuretic, history of syncope or severe unexplained faintness, known hypersensitivity to quinazolines
* Hemodynamically unstable
* Current use of over the counter, prescribed, or use of other drugs for insomnia
* Dependence on alcohol, opiates or other illegal drugs
* History of psychotic disorder
* Suicidal risk defined by a positive response on the 3-item assessment, standard protocol in the ED
* Current use of morphine or methadone
* Pregnant or breastfeeding
* Known hepatic dysfunction
* Cardiac or vascular history including coronary artery disease
* Narcolepsy
* History of sleep apnea
* Returning to chronic domestic abuse situation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Enrollment is limited to females for the purposes of limiting confounding factors in a small sample, and because many more females than males are treated for sexual assault.
Enrollment: 0 (Actual)
Dates: Start 2020-02-23 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptoms and severity - Clinician-Administered PTSD Scale - 5 (CAPS-5) | The full interview takes 45-60 minutes to administer and will be given at baseline, at approximately 31 days post event, and at three months.
  Clinician-Administered PTSD Scale-5 (CAPS-5) - Past Month & Past Week. The CAPS is the gold standard in PTSD assessment and the total score will serve as the primary outcome. The CAPS-5 is a 30-item structured interview to make a current (past month) diagnosis of PTSD, a lifetime diagnosis of PTSD, and assess PTSD symptoms over the past week. The full interview takes 45-60 minutes to administer and will be given at baseline, at approximately 31 days post event, and at three months.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | The PSQI will be completed weekly through study completion (average three months).
  The PSQI is a 19-item self-report questionnaire that assesses sleep quality over a 1-month interval. The questionnaire takes 10-15 minutes to complete. Total score from PSQI will be a secondary outcome of sleep with higher score indicating poorer sleep quality.
Pittsburgh Sleep Quality Index - Trauma Addendum (PSQI-A) | The PSQI-A will be completed weekly through study completion (average three months).
  The PSQI-A is a 7-item self-report questionnaire administered in conjunction with PSQI to examine the frequency of seven disruptive nocturnal behaviors common to PTSD among adults. Total score on PSQI-A will be a secondary outcome of trauma-associated sleep issues.
Patient Health Questionnaire (PHQ-9) | It takes about five minutes to complete and will be assessed weekly for the first seven weeks of participation and at three months/study completion (at each study visit).
  The PHQ-9 is a 10-item self-report questionnaire used in screening, diagnosing, monitoring, and measuring the severity of depression. Using an independent structured mental health professional interview as the criterion standard, a PHQ-9 score of 10 or more corresponded to good sensitivity and specificity (both 88%) for major depression.33 Total score will be a secondary outcome of depression symptom severity and score >=10 will be used to indicate major depression at 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873